CLINICAL TRIAL: NCT05272891
Title: The Effect of Audiobook Application on Anxiety, Depression and Quality of Life in Patients Receiving Hemodialysis Treatment
Brief Title: Audiobook Application in Patients Receiving Hemodialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Sevgi DEMIR CAM, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Sevgi Tez
Record Dates: First submitted 2022-02-04; First posted 2022-03-10 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Hemodialysis
Keywords: Anxiety; Depression; Quality of Life; nurse; Audio book
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: After determining the patients who meet the inclusion criteria, a randomization program will be used to ensure homogeneous distribution among the groups (Random Allocation Software). A list will be created according to the randomization program and 60 patients included in the study will be assigned to the experimental (30 patients) and control groups (30 patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): audio book will be played
  Interventions: Other: experimental group
- Control Group (No Intervention): No application will be made

INTERVENTIONS:
Other: experimental group — audio book app
  Other Names: experimental group, audio book app
  Arms: Experimental

SUMMARY:
This research will be conducted to evaluate the effects of audio book application on anxiety, depression and quality of life in patients receiving hemodialysis treatment.

DETAILED DESCRIPTION:
Hemodialysis is an extracorporeal blood purification technique used to remove accumulated metabolic waste products in patients and is a frequently used treatment method in patients with end-stage renal disease.

Although hemodialysis, which is one of the treatment of end-stage renal disease, prolongs life, it can also lead to various psychological disorders such as depression, anxiety and severe stress. Psychological disorders and depression in dialysis patients often manifest as a response to loss of ability to work and earn an income, decreased energy, decreased sexual function, other limitations caused by physical disability, and reduced life expectancy.

Depression is the most common psychopathological condition in patients with end-stage renal disease. The rate of depressive symptoms among dialysis patients is high and its prevalence is up to 43%, and it is stated that it has a significant effect on quality of life. The psychological and somatic effects of depression can complicate the course of the chronic disease.

Reading books is one of the tools to heal mental disorders. Some individuals cannot read on their own due to aging, poor eyesight, or lack of literacy. An audiobook is a recording of a book read by an author, actor, celebrity, or amateur. Audiobooks are recommended for their friendliness, comfort, and emotional impact. Audiobooks are recommended to increase the quality of life of individuals and to protect social health.

This research will be conducted to evaluate the effects of audio book application on anxiety, depression and quality of life in patients receiving hemodialysis treatment.

Patient information form, hospital anxiety depression scale, SF-36 quality of life scale will be used to collect research data.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Receiving hemodialysis treatment for six months or longer,
* Receiving hemodialysis treatment three times a week,
* No problem with the sense of hearing,
* Has no handicap in answering the questions physically and mentally,
* No verbal communication disability (hearing and speaking),
* Can understand Turkish,
* Not having been diagnosed with a mental illness,
* Patients willing to participate in the study will be recruited

Exclusion Criteria:

* Those who want to withdraw from the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The effect of audio book application on anxiety and depression in patients receiving hemodialysis treatment | At the end of 4 weeks
  Hospital anxiety and depression scale will be used. The lowest score that patients can get from the scale is 0, and the highest score is 21.
The effect of audio book application on quality of life in patients receiving hemodialysis treatment. | At the end of 4 weeks
  Short form 36 (SF-36) for quality of life scale will be used.Their scores range from 0-100. Scores are positively oriented. Increasing score indicates better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi DEMİR ÇAM, Phd Student, Principal Investigator — Ataturk University; Elanur YILMAZ KARABULUTLU, Prof.Dr., Study Director — Ataturk University
Locations (1):
- Hemodialysis units affiliated to Artvin provincial health directorate, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cam SD, Karabulutlu EY. Effects of Listening to an Audiobook on Anxiety, Depression, and Quality of Life in Patients Receiving Hemodialysis: A Randomized Controlled Trial. Hemodial Int. 2025 Oct;29(4):662-671. doi: 10.1111/hdi.13250. Epub 2025 May 29. PMID 40442032